CLINICAL TRIAL: NCT05530655
Title: A Phase I Study to Determine the Preferred Dose of the Angiotensin Converting Enzyme Inhibitor Lisinopril for Preventing Urinary Toxicity Following Radiotherapy for Prostate Cancer
Brief Title: A Study to Determine the Preferred Dose of the Drug, Lisinopril, for Preventing Urinary Toxicity Following Radiotherapy for Prostate Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Hong Zhang, Professor, University of Rochester
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007510_URGUP23077
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Radiation Toxicity; Urinary Complication
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries | interventions — Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients who receive radiation but no intervention
- Intervention group (Experimental)
  Interventions: Drug: Lisinopril Tablets

INTERVENTIONS:
Drug: Lisinopril Tablets — This is a dose escalation study of 5 mg, 10 mg and 20 mg doses given once a day.
  Arms: Intervention group

SUMMARY:
This study will establish the preferred dose of lisinopril in men with non-metastatic prostate cancer undergoing radiation treatment. This study will also evaluate the effect of lisinopril on urinary symptoms and the impact of lisinopril on biomarkers and their association with urinary symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of adenocarcinoma of the prostate and are candidates for curative-intent external beam radiation (with or without androgen deprivation therapy, ADT) at the Wilmot Cancer Institute Department of Radiation Oncology. Radiotherapy may be either primary, adjuvant or salvage. It may be part of combined treatment with androgen deprivation therapy.
* Be stage M0 based on the standard of care staging imaging
* Be able to read English
* Have the psychological ability and general health that permits completion of the study requirements and required follow up
* Be ≥18 and < 70 years of age
* Have ECOG performance status of 0 to 2 within 180 days prior to enrollment
* Have adequate renal function with creatinine clearance > 30 mL/min within 30 days prior to registration
* Have hematologic and hepatic function deemed adequate for planned treatment by the treating investigator within 90 days prior to registration, including:
* hemoglobin ≥9.0 g/dL, independent of transfusion and/or growth factors
* platelet count ≥100,000/µL independent of transfusion and/or growth factors
* Have a baseline systolic blood pressure of >130.

Exclusion Criteria:

* Have received prior pelvic radiotherapy
* Be taking lisinopril or other RAS modifying drug within two months prior to registration
* Have had a prior allergic reaction to lisinopril

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in Expanded Prostate Index Composite score | baseline to 12 months
  Patient reported outcomes capturing urinary symptoms will be collected using the Expanded Prostate Index Composite (EPIC) patient reported outcome questionnaire prior to radiation on the first day of treatment, weekly during radiation, and approximately 1 month, 3 months, 6 months, and 12 months after radiation. The EPIC bladder domain score will quantify patient reported urinary symptoms. The EPIC bladder domain consists of 12 items each scored on a Likert scale with an overall score transformed to a 0-100 scale. A higher score indicates worse outcome.
change in the percentage of patients with positive blood test in urine | baseline to 12 months
percentage of participants who achieve a dose of 20 mg | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmot Cancer Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No